CLINICAL TRIAL: NCT00899639
Title: Correlation of Oncotype Dx With Image Features and Molecular Characteristics of Breast Cancer
Brief Title: Studying Tumor Tissue Samples From Patients With Early-Stage Breast Cancer
Status: Withdrawn | Type: Observational
Why Stopped: not "applicable clinical trial"
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: 000809; P30CA072720 (NIH); CDR0000600231; CINJ-0220080120
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; estrogen receptor-positive breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at tumor tissue samples from patients with early-stage breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To characterize differences in tumor morphology and molecular features that exist in good- and poor-prognosis breast cancer as determined by Oncotype Dx assay (a reverse transcriptase-PCR-based assay).
* To develop a computer-aided design (CAD)-based system of analysis of digitized histological images that would perform as well as Oncotype Dx assay in stratifying estrogen receptor-positive (ER+) breast cancer into prognostic categories.
* To identify new therapeutic targets in the PI3-kinase signaling pathway for a subset of poor-prognosis ER+ breast cancers.

OUTLINE: Patients who had Oncotype Dx assay (a reverse transcriptase-PCR-based assay) performed for their breast cancer are identified by review of medical records. Diagnostic H&E stained tumor tissue samples are reviewed by a pathologist. Relevant pathologic features of the tumor (size, stage, grade, estrogen receptor, progesterone receptor, and HER2 staining) and linked Oncotype Dx score are recorded.

The H&E stained tumor tissue samples are scanned to create high-resolution digital images. The images from each tissue sample are subjected to image analysis algorithms to identify sets of image features that most clearly separate tumors with low recurrence scores from those with high recurrence scores.

Unstained paraffin sections from each tumor tissue sample, when available, are processed using IHC to analyze PI3-kinase signaling pathway (PTEN expression). Staining for other components of the PI3-kinase signaling pathway, phospo-AKT, and other proteins of interest is also performed. DNA is extracted from the samples and subjected to pyrosequencing analysis on exons 9 and 20 of PI3KCA. Sequencing of other relevant potential oncogenes, such as AKT, is also performed. Statistical analysis is performed to look for a correlation between Oncotype Dx scores and the presence of PI3KCA mutations and/or loss of PTEN expression.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of early-stage breast cancer for which an Oncotype Dx assay has been performed
* Must have diagnostic H&E stained tumor tissue samples available
* Hormone receptor status:

  * Estrogen receptor-positive tumor

PATIENT CHARACTERISTICS:

* Menopausal status not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ER+ breast cancer with associated Oncotype Dx scores
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-05; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Differences in tumor morphology and molecular features that exist in good- and poor-prognosis breast cancer as determined by Oncotype Dx assay
Histological image-based analysis in stratifying estrogen receptor-positive breast cancer into prognostic categories
Identification of new therapeutic targets in the PI3-kinase signaling pathway for a subset of poor-prognosis estrogen receptor-positive breast cancers

CONTACTS AND LOCATIONS:
Overall Officials: Shridar Ganesan, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey